CLINICAL TRIAL: NCT04829084
Title: Augmenting the Referral Pathway to Improve the Uptake of Retinal Services Among Diabetic Patients at Reiyukai Eiko Masunaga Eye Hospital, Nepal, a Non-randomized Pre-post Intervention Study
Brief Title: Augmenting Referral Pathway to Improve Uptake of Retinal Services by Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seva Foundation (Other)
Collaborators: Reiyukai Eiko Masunaga Eye Hospital (REMEH) (Unknown); Indian Institute of Public Health, India (Other); Seva Canada Society (Other); Queen's University, Belfast (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: REMEH/ERB/582/2020 P
Record Dates: First submitted 2021-03-30; First posted 2021-04-02 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetes; Diabetic retinopathy; Nepal; Health education; Referral
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus; Health Education

STUDY DESIGN:
Intervention Model Description: To Increase the attendance of patients with Diabetes Mellitus, for retinal screening at REMEH by providing health education intervention to selected physicians and establishing a referral pathway.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Health education
  Interventions: Behavioral: Pre-post educational intervention
- Control Arm (No Intervention): No health education

INTERVENTIONS:
Behavioral: Pre-post educational intervention — To Increase the attendance of patients with Diabetes Mellitus, for retinal screening at REMEH by providing health education intervention to selected physicians and establishing a referral pathway
  Arms: Intervention Arm

SUMMARY:
Reiyukai Eiko Masunaga Eye Hospital (REMEH) is a non-profitable organization. Retina services were resumed from October 2019. Until this retinal service started, it has been mostly cataract-focused. People are unaware of this new retinal service in the hospital. The investigators would like to fill this gap and our objective is to increase the attendance of patients with Diabetes Mellitus, for retinal screening at REMEH by providing health education intervention to selected physicians and establish a referral pathway.

Study Design: pre- post-intervention Methods: The investigators are going to conduct intervention by providing health education on diabetes Retinopathy to the health personnel of Scheer Memorial Hospital. It has been referring eye patients to REMEH as there is no eye department there.

Data Management: The demographic information of health personnel of Sheer memorial and demographic information and other variables of the patient who are referred from Scheer Hospital will be collected and entered in an excel sheet.

The study period of approximately 16 months (March 2020 to Sep 2021): Initial 10 months for proposal writing, preparation, and getting ethical approval. Feb2021 - April 2021 three months for pretest intervention May- July further data collection and last two months Aug- Sep Analysis and writing result.

Results: The proposed outcome is to increase the proportional change in the number of patients availing retinal services and to find out a proportional increase in the number of diabetes screenings from the baseline. Also, a positive outcome is a clear indication for health education, and setting communication between general physicians and specialties will set the path for improvement in a timely health care delivery system.

DETAILED DESCRIPTION:
Diabetes Mellitus (DM) is a chronic, metabolic disease characterized by elevated levels of blood glucose (or blood sugar), which leads over time to serious damage to the heart, blood vessels, eyes, kidneys, and nerves. People with diabetes can develop an eye disease called Diabetic Retinopathy when high blood sugar levels damage the blood vessels in the retina. Diabetic Retinopathy if detected early can be treated to preserve the vision. Once the vision has been lost it cannot usually be restored. Diabetic retinopathy is an emerging cause of blindness in developing countries. Diabetic retinopathy is a common and specific microvascular complication of diabetes and remains the leading cause of preventable blindness in working-aged people. It is identified in a third of people with diabetes and associated with an increased risk of life-threatening systemic vascular complications, including stroke, coronary heart disease, and heart failure.

The worldwide prevalence of diabetic retinopathy (DR) was found to be 34.6%. WHO estimates that DR is responsible for 4.8% of the 37 million cases of blindness throughout the world. Diabetic retinopathy (DR) is the fifth leading cause of visual impairment and the fourth leading cause of blindness in the world (WHO, TADDS). In a study undertaken in an urban population in Nepal, M.D.Bhattarai found the prevalence of diabetes among people aged 20 years and above to be 14.6% and the prevalence among people aged 40 years and above to be 19%. KAP study in Kathmandu revealed good knowledge, good attitude but poor practice among the diabetic group. In contrast, the non-diabetic groups showed poor knowledge but a good attitude and poor lifestyle practices. Hence diabetic group needs good practice like early diagnosis of DR and self-care, and the non-diabetic group needs knowledge. Simply increasing awareness among diabetic patients about the risk factors is not sufficient to improve ophthalmic care. Various strategies will be necessary to improve good practice and patient visits to an eye clinic on a regular basis.

Reiyukai Eiko Masunaga Eye Hospital (REMEH) was established in February 2007. REMEH is a non-profitable organization. Approximately 411,057 populations of Kavrepalanchowk district are the catchment area of REMEH. The REMEH hospital provided OPD service to 43,787 patients in 2018 and 54,213 patients in 2019, performed 1,058 cataract surgeries in 2018 and 1,647 in 2019. Similarly, retina services were resumed from October 2019.

People are unaware of this new retinal service in the hospital. There was irregular retinal service due to the lack of a vitreoretinal surgeon. But now there is regular medical as well as surgical retina service. The unavailability of retina surgeons, low literacy rate and the lack of awareness programs conducted in the community, costly retinal services, lack of proper linkage to diabetic clinics and REMEH could be a reason for the low uptake of retina services. The investigators would like to fill this gap and increase the uptake of this retina sub-specialty focusing on Diabetes Mellitus to decrease blindness caused by Diabetic Retinopathy by augmenting the referral pathway and declining the problem tree.

Methods:

This study is operational research that will take place in REMEH. The study design is a non-randomized pre and post-intervention study design without a control group. The intervention will consist of Health Education to specific health personnel who deal with DM patients. A multi-specialty hospital named Scheer Memorial Hospital will be the intervention hospital. Through the intervention, a referral pathway will be created to send the diabetes patients for diabetic retinopathy screening to REMEH.

Research Objective:

Primary Objective: To provide health education intervention to selected health personnel and establish a referral pathway.

Secondary Objective: To increase the attendance of patients with Diabetes Mellitus for retinal screening at REMEH.

Details of the intervention hospital:

Scheer memorial hospital is a 150-bed hospital with daily 475 outpatient department patients. It is located 1.8 km away from REMEH and has 223 staff.

Intervention:

Using the complete enumerations of all health personnel treating patients with diabetes, below mentioned personnel will have more chances to interact with diabetic patients so only a total of 19 health personnel will be chosen. They are 4 physicians, 4 pediatricians, 8 medical officers, and 3 assistants of Scheer Hospital.

Actions expected from selected health personnel in Scheer Memorial

1. Counsel DM patients to visit REMEH
2. Use referral slip while referring patients to REMEH
3. Handover DR-related pamphlet to DM patients.

1. Record total cases referred to REMEH in a month Depending on the feasibility, the Pilot may be conducted with another group of doctors, to see if the materials are well understood and the duration is optimal. A pilot test will help to see the smoothness of the sessions conducted. Necessary modification in the PPT, method of training delivery if needed will be done for the training sessions after the pilot Pilot visit: It will include the same IEC materials used for intervention. PPT presentation by retina specialist with ample time to answer queries. One short video display. Distribution of posters, pamphlets,

1. st visit: The information sheet with the consent form will be shared. The pre-test will be done. PPT presentation by retina specialist with information on DR and importance of the timely visit to screen eyes for DM patients will be presented. Distribution of posters, pamphlets will be done.
2. nd visit: Two video presentations about Diabetic Retinopathy will be done. And posters and pamphlets will be distributed.
3. rd visit: Refresher of previous sessions. A small quiz about the knowledge about DR among the health personnel will be done and a post-test will be done about the acquired knowledge.

Data collection:

Baseline data collection has been started from 1st June 2020 and has been continued till 25th February 2021.

Time Management for the manuscript-

1. Preparation (three months: March 2020 to December 2020) The first 10 months will be used for planning, proposal writing, and getting ethical approval from Nepal Health Research Council. Scheer Memorial will be requested for approval of the study.
2. Pre-test and Intervention (February 2021 to April 2021) Baseline data will be collected from June 1st to February 25th and the intervention started on 26th February 2021. Initially, the Scheer Memorial hospital will be visited by the management team and the procedure regarding the project will be explained including the patient referral process. Similarly, a register will be maintained at REMEH to get demographic information of each and every Diabetes Mellitus patient and information on the referral physician/hospitals or self-referral visiting REMEH. Monthly data will be collected from both the hospital regarding the number of patients referred for DR screening. Pretest to see the smoothness of the training will be done and then monthly once visits will be done at Scheer Memorial for intervention.
3. Data collection (Four months: May 2021 to July 2021) The data will be collected for another three months ie: May to July 2021. Data on demographic detail of health personnel, pre, and post-test scoring will be collected. Data on demographic details, referral hospital, presence and stage of DR, visual outcome of patients will also be collected.
4. Data analysis and Manuscript writing: (2 months: August- September 2021) The last 2 months August and September will be for data analysis and manuscript writing.

Study Subjects:

Target population: Health care personnel Study participants: Selected health care personnel from Scheer Memorial Hospital hospital.

Sampling techniques: Complete enumerations of all health personnel treating diabetic patients.

The procedure of Data Collection: Primary data collection will be done by a single person who assists in OPD and who will be designated for data collection. The register will be maintained at REMEH and monthly data on the number of DM patients referred for DR screening will be collected from Scheer Memorial. These data will later be entered into Microsoft Excel files or SPSS on weekly basis.

Project Strategies /Activities and patient pathway:

The study will be explained to Scheer Memorial Hospital

* Intervention in Scheer Memorial Hospital to do awareness campaigns and refer diabetic patients to REMEH.
* The health personals will be acknowledged in the study.
* A referral slip/ written communication will be made and the referral process will be a vice versa feedback process.
* Screening of all Diabetes patients will be done at REMEH by dilated fundus examination under slit-lamp biomicroscopy.
* Dilated fundus examination of diabetic patients visiting the hospital will be done by slit-lamp biomicroscopy.

When the participants enter REMEH for retinal services firstly the patient will be assessed. The demographic data along with the referred physician or self-referral will be noted. It will include history focused on diabetes and its modifiers. History of patients includes: duration of diabetes, past glycemic control (hemoglobin A,1c), Medications (especially insulin, oral hypoglycemic, anti-hypertensives, and lipid-lowering drugs), mention whether simply diet control or herbal, systemic history (e.g., renal disease, systemic hypertension, serum lipid levels, pregnancy, Anemia, Cardiac condition), ocular history smoking history and contact information.

The screening will be made according to WHO tools for assessment of Diabetic Retinopathy. Detailed patient assessment will include a complete ophthalmic examination, including visual acuity and the identification and grading of severity of DR and presence of DME for each eye.

Physical examination of the eye will include: Visual acuity, measurement of intraocular pressure (IOP), gonioscopy when indicated (e.g., when neovascularization of the iris is seen or in eyes with increased IOP), slit-lamp bio-microscopy for anterior segment evaluation, and fundus examination.

The follow-up will be scheduled according to the National Guidelines for Management of Diabetic Retinopathy 2017.

Data entry and Analysis: Data entry and management will be done by the optometrist. Statistical Package for the Social Sciences (SPSS) version 20 will be used in the end just before project outcomes.

Ethical approvals: Ethical approval taken from Nepal Health Research Council (NHRC)

Discussion:

Our study is a non-randomized pre and post-intervention design which includes the collaboration between an eye hospital and multi-specialty hospital focusing on the health professional as a stakeholder to increase the referral of diabetic. The stakeholders will be provided health education on awareness of diabetic retinopathy using PPTs, posters, pamphlets, and referral slips. The outcome of the intervention will be assessed by a pre-and post-evaluation questionnaire.

There are few studies similar to ours that have assessed the awareness of physicians by calculating the Diabetic retinopathy awareness index. Anwar et al conducted a 27-item consented & validated, multiple-choice questionnaire based on physician's characteristics, knowledge, and practice of diabetic eye care and challenges faced due to the current DR referral system in Pakistan.

The investigators will use a referral slip as a mode of communication between an ophthalmologist and health care personnel with reference to the referral of diabetic patients. Storey et al found that written communication between an ophthalmologist and a primary care physician (PCP) and referral vice versa was effective to change the behavior of the referring physicians. Riordan et al assessed that phone /letter reminder to patient and provider level training increased diabetic screening. Printed educational messages or posters also increased behavior and attitude change to primary care physicians.

Grimshaw et al also found that printed educational messages increased the number of referrals by primary care physicians similar to our study where the investigators are using referral slips to communicate between the ophthalmologist and health Health education intervention could be a low-cost solution to improve the awareness, access, utilization of retinal health care services; thus, health education intervention could reduce the burden of DR among people with diabetes. However, this is an unexplored area in Nepal. Working closely with the stakeholders, this study will evaluate the role of health education interventions (which are already validated in other low-income settings) to reduce the burden of DR in Nepal.

Strength and Limitations:

The strength of our study is that it will be one of the first studies including stakeholders to increase the attendance of diabetic retinopathy in Nepal. This helps to reduce the unavoidable blindness caused by diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Complete enumerations of all Health Personnel treating patients with Diabetes.

Exclusion Criteria:

* Health Personnel who are not directly linked with treating patients with Diabetes.
* Health personnel not willing to participate in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Increased number of DR patients at REMEH for eye screening | 4 months
  The proposed result of the study is the proportional change in number of patients availing retinal services will be calculated and to find out proportional increase in number of diabetes screening from the baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Reiyukai Eiko Masunaga Eye Hospital (REMEH), Banepa, Nepal

REFERENCES:
- [Derived] Shrestha R, Singh P, Dhakwa P, Tetali S, Batchu T, Thapa PS, Agiwal V, Pant H. "Augmenting the referral pathway for retinal services among diabetic patients at Reiyukai Eiko Masunaga Eye Hospital, Nepal: a non-randomized, pre-post intervention study". BMC Health Serv Res. 2023 Feb 8;23(1):126. doi: 10.1186/s12913-023-09105-3. PMID 36750897
- [Derived] Shrestha R, Singh P, Dhakhwa P, Tetali S, Batchu T, Shrestha Thapa P. Augmenting the Referral Pathway for Retinal Services Among Patients With Diabetes Mellitus at Reiyukai Eiko Masunaga Eye Hospital, Nepal: Protocol for a Nonrandomized, Pre-Post Intervention Study. JMIR Res Protoc. 2021 Dec 17;10(12):e33116. doi: 10.2196/33116. PMID 34927596